CLINICAL TRIAL: NCT04034277
Title: Lee Silverman Voice Treatment Versus Standard Speech and Language Therapy Versus Control in Multiple Sclerosis: a Randomized Controlled Trial
Brief Title: Lee Silverman Voice Treatment Versus Standard Speech Therapy Versus Control in Hypophonia Rehabilitation in MS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Davide Cattaneo, Research Coordinator Larice Lab., Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SM_Voice_RCT
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Multiple Sclerosis
Keywords: Voice Disorders; Speech and language therapy; Lee Silverman voice treatment
MeSH Terms: conditions — Multiple Sclerosis; Voice Disorders; Communication Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lee Silverman Voice Therapy (Experimental): LSVT LOUD® is a therapy program which requires four sessions per week for 4 weeks by a speech and language therapists with a certification in Lee Silverman Voice Therapy. Each session lasted 50-60 min.
  Interventions: Other: Lee Silverman Voice Therapy
- Conventional Treatment (Active Comparator): The content and dose of standard SLT is poorly defined within the published literature. For this reason, the standard therapy intervention will encompass all SLT techniques that are not LSVT®. Treatment will be individualized and may include any of the following: exercises targeting respiration, phonation, articulation, behavioral strategies to reduce prosodic abnormality
  Interventions: Other: Conventional Treatment

INTERVENTIONS:
Other: Lee Silverman Voice Therapy — LSVT LOUD® comprises maximum effort non-speech and speech drills. The non-speech drills include the production of 15 sustained 'ah' phonation at high volume and pitch glides (5 repetitions moving from modal pitch to high pitch and 15 repetitions moving from modal pitch and going down on production of sustained 'ah'). The speech drills utilize a hierarchy of speech tasks moving from single words through phrases and onto conversational speech to generalize
  Arms: Lee Silverman Voice Therapy
Other: Conventional Treatment — speech rehabilitation protocol comprehend:
  * Respiratory and phonatory exercises: exercises to increase diaphragmatic and respiratory functions, exercises to increase expiration time using natural expiration or sibilant, exercise to increase phonation time by pronouncing the vocal /a/, exercise to reduce oral stiffness.
  * Articulation and prosody exercises: repetition or reading lists of possibly long and complex words that start with or contain consonants groups. Read aloud texts, sentences or words, making sure to articulate and pronounce the words well without diminishing or increasing the rhythm of speech, with the correct punctuation and intonation. If necessary, ask patients to hyperarticulate, accelerate or slow down, or exaggerate intonation.
  Arms: Conventional Treatment

SUMMARY:
The aim of the study is to identify the most effective method of intervention to reduce hypophonia in PwMS (Patient With Multiple Sclerosis), as a way to optimize the speech-therapy treatment based on scientific evidence. In the previous AB study, we aimed to verify the efficacy of LSVT LOUD® in PwSM: in the present study we will compare different treatment in a larger sample.

Half of the participants will follow the LSVT Loud program, the other half will follow usual care rehabilitation programs.

The results of these groups will be compared with an historical cohort of no treatment patients.

DETAILED DESCRIPTION:
The descriptive studies showed that voice problems, in particular hypophonia, are present in 45% to 91% of patients with multiple sclerosis and may constitute a limitation in social life participation. Although voice, speech and communication are significant aspects for the biopsychosocialwell-being and life quality, only 2% of the PwMS had received any speech therapy and, at the same time, few studies assessed the effects of speech treatment for PwMS.

In according to the taxonomy of voice therapy, the conventional treatment may include direct interventions such as vocal function and modification of respiratory function.

The LSVT LOUD® treatment is a standardized, research-based speech treatment protocol with established efficacy for Idiopathic Parkinson Disease (IPD) and is well described in a large number of studies. Subsequently, further studies supported the efficacy of LSVT LOUD® in voice rehabilitation in various neurological diseases, including Multiple Sclerosis. In the study of Sapir et al., only two women were treated with LSVT LOUD® and the authors concluded that intensive phonatory-respiratory treatment can produce clinically significant and long-term improvement in vocal function in PwMS. These findings are consistent with suggestion that intensive training can improve function in those parts of the body that are prone to fatigue and that vocal training probably minimizes disuse atrophy and increases muscle strength and coordination.

The content and dose of the SLT (Speech Language Therapy) of dysphonia in MS is poorly defined within the published literature and we did not find any meta-analyzes or guidelines that suggest instructions for therapists.

The purpose of this project is to identify the most effective method of intervention to reduce hypophonia in PwMS, as a way to optimize the speech-therapy treatment based on scientific evidence. The data in literature suggest that LSVT LOUD® may be functional for these aims, although there isn't broad-based study with PwSM.

Fourty Persons with Multiple Sclerosis will be randomly allocated to an experimental group (Lee Silverman Voice Treatment - LSVT LOUD® method) or to a control group following usual care rehabilitation programs.

Also an historical cohort of untreated patients was considered (voice assessment: baseline, after 4 weeks, FU-Follow Up at 6/12 months).

Data collection in both groups will be performed at baseline, after 4 weeks of treatment and after 6-12 months up to the end of the rehabilitation program (FU). In order to evaluate the perceptual impact of the treatment, GIRBAS and VHI will be proposed.

The acoustic variables will be recorded with the software PRAAT: SPL (Sound Pressure Level) of a sustained /ah/, SPL of functional sentences, maximum phonation time, SPL of 1 minute monologue. In addition, the following values were taken in the minute of spontaneous speech: Jitter, shimmer, fundamental frequency, maximum frequency and minimum frequency. The type of MS, Expanded Disability Status Scale (EDSS) , demographic data, disease duration, presence of postural and respiratory problems, presence of depression (Beck Depression Inventory-II - BDI II) , pharmacological treatment and cognitive status (Brief Repeatable Battery of Neuropsychological Tests) will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Sclerosis according with McDonald's criteria;
* absence of relaps in the last month;
* Mini Mental State Examination (MMSE) > 21 score for a better understanding and adherence to the execution of the proposed exercises;
* hypophonia (conversation < 60 dB SPL- distance was kept equal at about 15 cm);
* ability to understand the aims of the study and acceptance to sign an informed consent;
* acceptance of the intensity of the treatment;
* ability to understand the Italian language.

Exclusion Criteria:

* Presence of other neurological disorders;
* visual/hearing impairments hindering the rehabilitation program;
* clinical history of laryngeal cancer, chemotherapy, radiotherapy, head and neck trauma or endotracheal intubation;
* relapse or sudden changes in their MS symptoms within the previous 3 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in intensity (dB) of 3 sustained /ah/ | at baseline, at 4 weeks (after the completion of 16 training sessions) and after 6-12 months up to the end of the rehabilitation program (FU)
  All subjects were requested to sustain the vowel /ah/ as long as possible at a comfortable frequency and maximum intensity level. Specific task was given: "Please and say /ah/. Make it strong and steady, and sustain it for as long as you can".
Change in intensity measured in decibel (dB) of three functional sentences | at baseline, at 4 weeks (after the completion of 16 training sessions) and after 6-12 months up to the end of the rehabilitation program (FU)
  all speakers were requested to produce three functional sentences at a comfortable frequency and maximum intensity level. The sentences were the same for all subjects. Specific tasks, identical for each individual, was given: "Please take a deep breath and repeat each sentences with effort voice".
Change in intensity in conversation measured in decibel (dB) | at baseline, at 4 weeks (after the completion of 16 training sessions) and after 6-12 months up to the end of the rehabilitation program (FU)
  A speech sample of approximately one minute of spontaneous conversation was recorded and measured in dB in order to analyze speech intensity. Specific tasks, identical for each individual, was given: "Please speak for at least a minute".

SECONDARY OUTCOMES:
Change in Maximum Phonation Time (MPT) of three sustained /ah/ (sec.) | at baseline, at 4 weeks (after the completion of 16 training sessions) and after 6-12 months up to the end of the rehabilitation program (FU)
  All subjects were requested to sustain the vowel /ah/ as long as possible at a comfortable frequency and maximum intensity level. Specific tasks, identical for each individual, was given: "Please and say /ah/. Make it strong and steady, and sustain it for as long as you can".
Change in Vocal Handicap Index | at baseline, at 4 weeks (after the completion of 16 training sessions) and after 6-12 months up to the end of the rehabilitation program (FU)
  Voice Handicap Index (VHI) is a self-assessed standardized 30-point questionnaire, which includes items on the impact of the voice disorder on daily life. The questionnaire is divided into three subscales covering functional, emotional and physical aspect of voice disorders. Each answer is graded 0 to 4 depending on the frequency of the difficulty: 0 no difficulties, 1 almost never, 2 sometimes, 3 almost always, 4 always.
Change in GIRBAS | at baseline, at 4 weeks (after the completion of 16 training sessions) and after 6-12 months up to the end of the rehabilitation program (FU)
  Tool used to quantify perceptual evaluation of the voice quality. The scale evaluates in particular 5 aspects of voice: Grade, Instability, Roughness, Breathiness, Asthenia, and Strain. Voice quality was assessed by a trained speech therapist, using a scale from 0 to 3 where 0 regular, 1 mildly pronounced, 2 moderate, 3 very pronounced.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Carrozza, PhD, Study Director — Fondazione Don C. Gnocchi
Locations (1):
- Fondazione Don Gnocchi Irccs, Milan, Italy